CLINICAL TRIAL: NCT01040572
Title: Laparoscopic Revision Gastric Bypass Surgery for Weight Recidivism: Our Experience in 170 Patients
Brief Title: Laparoscopic Revision Gastric Bypass for Weight Recidivism
Acronym: WR
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D. Higa, MD; FACS; FASMBS; Clinical Professor of Surgery, UCSF, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2009078; U1111-1113-0216 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-23; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-10

CONDITIONS: Weight Regain; Weight Recidivism; Obesity Recidivism; Clinically Severe Obesity
Keywords: Obesity recidivism; Weight Regain; Weight recidivism; Morbidity; Complication; Late complications; Revisional gastric bypass; Re-operative gastric bypass; Revisional bariatric surgery; Re-operative bariatric surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obesity recidivism after gastric bypass

SUMMARY:
The main aim of this study is to analyze and report traditional, patient-centered, and composite intermediate-term outcomes after laparoscopic revision Roux-en-Y gastric bypass surgery for weight recidivism.

DETAILED DESCRIPTION:
There is lack of standardization of primary and revisional bariatric surgery compounded by a scant long-term outcome data. The treatment of inadequate weight loss, weight recidivism, and most severe technical complications after primary bariatric surgery remains refractory to non-operative treatment. Failure rates have been reported up to 20% and 35% for the morbidly obese (MO) and super obese (SO), respectively at 2 to 3 years after surgery. The indication for further surgical intervention remains controversial, as does what type of revisional procedure, both operative and endoscopic, to recommend. Furthermore, there is no standardization of the limb lengths, pouch size or the use of prosthetic reinforcement. Therefore the approach to these patients must be as individualized as their original operations. We formally analyze our experience with all laparoscopic revisional strategies for weigh regain after failed gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent laparoscopic revisional "RYGB" for failed "RYGB" with weight recidivism or weight regain "WR" pattern

Exclusion Criteria:

* failed RYGB with an Inadequate Initial Weight Loss "IIWL" pattern
* patients with prior major bariatric conversion or esophago-gastric surgeries
* RYGB patients revised by an open surgical approach
* RYGB patients who underwent laparoscopic revisional RYGB surgery somewhere else and continue their follow-up care with our program
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously failed Roux-en-Y gastric bypass "RYGB" surgery with a weight recidivism pattern.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight loss expressed as Body Mass Index and Percentage Excess Weight Loss | At the lowest weight loss point and at last follow-up
Comorbidity status | throughout follow-up
Subjective Satisfaction | at last follow-up
Health-Related Quality of Life (HR-QoL). | at the last follow-up
Morbidity and mortality | throughout follow-up

SECONDARY OUTCOMES:
To assess failures | at yearly intervals throughout follow-up
To evaluate the patients´ metabolic and nutritional status | throughout follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- UCSF Fresno Center for Medical Education and Research, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Calle EE, Thun MJ, Petrelli JM, Rodriguez C, Heath CW Jr. Body-mass index and mortality in a prospective cohort of U.S. adults. N Engl J Med. 1999 Oct 7;341(15):1097-105. doi: 10.1056/NEJM199910073411501. PMID 10511607
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] www.asbs.org/htm/Private/resolution.html. American Society for Metabolic and Bariatric Surgery.
- [Background] O'Brien PE, McPhail T, Chaston TB, Dixon JB. Systematic review of medium-term weight loss after bariatric operations. Obes Surg. 2006 Aug;16(8):1032-40. doi: 10.1381/096089206778026316. PMID 16901357
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Ann Surg. 2006 Nov;244(5):734-40. doi: 10.1097/01.sla.0000217592.04061.d5. PMID 17060766
- [Background] Sarr MG. Reoperative bariatric surgery. Surg Endosc. 2007 Nov;21(11):1909-13. doi: 10.1007/s00464-007-9536-x. Epub 2007 Aug 19. No abstract available. PMID 17705073
- [Background] Schwartz RW, Strodel WE, Simpson WS, Griffen WO Jr. Gastric bypass revision: lessons learned from 920 cases. Surgery. 1988 Oct;104(4):806-12. PMID 3051478
- [Background] Khaitan L, Van Sickle K, Gonzalez R, Lin E, Ramshaw B, Smith CD. Laparoscopic revision of bariatric procedures: is it feasible? Am Surg. 2005 Jan;71(1):6-10; discussion 10-2. PMID 15757050
- [Background] Roberts K, Duffy A, Kaufman J, Burrell M, Dziura J, Bell R. Size matters: gastric pouch size correlates with weight loss after laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2007 Aug;21(8):1397-402. doi: 10.1007/s00464-007-9232-x. Epub 2007 Mar 1. PMID 17332953
- [Background] Madan AK, Tichansky DS, Phillips JC. Does pouch size matter? Obes Surg. 2007 Mar;17(3):317-20. doi: 10.1007/s11695-007-9058-6. PMID 17546838
- [Background] Muller MK, Wildi S, Scholz T, Clavien PA, Weber M. Laparoscopic pouch resizing and redo of gastro-jejunal anastomosis for pouch dilatation following gastric bypass. Obes Surg. 2005 Sep;15(8):1089-95. doi: 10.1381/0960892055002257. PMID 16197777
- [Background] Patel RA, Brolin RE, Gandhi A. Revisional operations for marginal ulcer after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2009 May-Jun;5(3):317-22. doi: 10.1016/j.soard.2008.10.011. Epub 2008 Nov 6. PMID 19136312
- [Background] Fobi MA, Lee H, Felahy B, Che K, Ako P, Fobi N. Choosing an operation for weight control, and the transected banded gastric bypass. Obes Surg. 2005 Jan;15(1):114-21. doi: 10.1381/0960892052993404. PMID 15760509
- [Background] Capella JF, Capella RF. An assessment of vertical banded gastroplasty-Roux-en-Y gastric bypass for the treatment of morbid obesity. Am J Surg. 2002 Feb;183(2):117-23. doi: 10.1016/s0002-9610(01)00871-6. PMID 11918873
- [Background] White S, Brooks E, Jurikova L, Stubbs RS. Long-term outcomes after gastric bypass. Obes Surg. 2005 Feb;15(2):155-63. doi: 10.1381/0960892053268282. PMID 15802056
- [Background] Bessler M, Daud A, Kim T, DiGiorgi M. Prospective randomized trial of banded versus nonbanded gastric bypass for the super obese: early results. Surg Obes Relat Dis. 2007 Jul-Aug;3(4):480-4; discussion 484-5. doi: 10.1016/j.soard.2007.01.010. Epub 2007 Jun 4. PMID 17544335
- [Background] Z'graggen K, Guweidhi A, Steffen R, Potoczna N, Biral R, Walther F, Komminoth P, Horber F. Severe recurrent hypoglycemia after gastric bypass surgery. Obes Surg. 2008 Aug;18(8):981-8. doi: 10.1007/s11695-008-9480-4. Epub 2008 Apr 26. PMID 18438618
- [Background] Dapri G, Cadiere GB, Himpens J. Laparoscopic placement of non-adjustable silicone ring for weight regain after Roux-en-Y gastric bypass. Obes Surg. 2009 May;19(5):650-4. doi: 10.1007/s11695-009-9807-9. Epub 2009 Mar 5. PMID 19263180
- [Background] Kyzer S, Raziel A, Landau O, Matz A, Charuzi I. Use of adjustable silicone gastric banding for revision of failed gastric bariatric operations. Obes Surg. 2001 Feb;11(1):66-9. doi: 10.1381/096089201321454132. PMID 11361171
- [Background] Bessler M, Daud A, DiGiorgi MF, Olivero-Rivera L, Davis D. Adjustable gastric banding as a revisional bariatric procedure after failed gastric bypass. Obes Surg. 2005 Nov-Dec;15(10):1443-8. doi: 10.1381/096089205774859173. PMID 16354525
- [Background] Gobble RM, Parikh MS, Greives MR, Ren CJ, Fielding GA. Gastric banding as a salvage procedure for patients with weight loss failure after Roux-en-Y gastric bypass. Surg Endosc. 2008 Apr;22(4):1019-22. doi: 10.1007/s00464-007-9609-x. Epub 2007 Oct 18. PMID 17943353
- [Background] Chin PL, Ali M, Francis K, LePort PC. Adjustable gastric band placed around gastric bypass pouch as revision operation for failed gastric bypass. Surg Obes Relat Dis. 2009 Jan-Feb;5(1):38-42. doi: 10.1016/j.soard.2008.08.012. Epub 2008 Aug 22. PMID 18996754
- [Background] Mouiel J, Bourg S, Iannelli A, et al. Nouvelle technique de gastroplatie verticale calibree type Mason-MacLean aveccure de reflux gastro-oesophagien. Jornal de Coelio Chirurgie 2001; 38: 53-6.
- [Background] Fedenko V, Evdoshenko V. Antireflux sleeve gastroplasty: description of a novel technique. Obes Surg. 2007 Jun;17(6):820-4. doi: 10.1007/s11695-007-9124-0. PMID 17879584
- [Background] Brolin RE, Kenler HA, Gorman JH, Cody RP. Long-limb gastric bypass in the superobese. A prospective randomized study. Ann Surg. 1992 Apr;215(4):387-95. doi: 10.1097/00000658-199204000-00014. PMID 1558421
- [Background] MacLean LD, Rhode BM, Nohr CW. Long- or short-limb gastric bypass? J Gastrointest Surg. 2001 Sep-Oct;5(5):525-30. doi: 10.1016/s1091-255x(01)80091-3. PMID 11986004
- [Background] Choban PS, Flancbaum L. The effect of Roux limb lengths on outcome after Roux-en-Y gastric bypass: a prospective, randomized clinical trial. Obes Surg. 2002 Aug;12(4):540-5. doi: 10.1381/096089202762252316. PMID 12194548
- [Background] Lee S, Sahagian KG, Schriver JP. Relationship between varying Roux limb lengths and weight loss in gastric bypass. Curr Surg. 2006 Jul-Aug;63(4):259-63. doi: 10.1016/j.cursur.2006.05.001. PMID 16843777
- [Background] Ciovica R, Takata M, Vittinghoff E, Lin F, Posselt AM, Rabl C, Stein HJ, Campos GM. The impact of roux limb length on weight loss after gastric bypass. Obes Surg. 2008 Jan;18(1):5-10. doi: 10.1007/s11695-007-9312-y. Epub 2007 Dec 7. PMID 18064526
- [Background] Bruder SJ, Freeman JB, Brazeau-Gravelle P. Lengthening the Roux-Y Limb Increases Weight Loss after Gastric Bypass: a preliminary report. Obes Surg. 1991 Mar;1(1):73-77. doi: 10.1381/096089291765561501. PMID 10715665
- [Background] Freeman JB, Kotlarewsky M, Phoenix C. Weight loss after extended gastric bypass. Obes Surg. 1997 Aug;7(4):337-44. doi: 10.1381/096089297765555593. PMID 9730521
- [Background] Feng JJ, Gagner M, Pomp A, Korgaonkar NM, Jacob BP, Chu CA, Voellinger DC, Quinn T, Herron DM, Inabnet WB. Effect of standard vs extended Roux limb length on weight loss outcomes after laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2003 Jul;17(7):1055-60. doi: 10.1007/s00464-002-8933-4. Epub 2003 May 6. PMID 12728380
- [Background] Inabnet WB, Quinn T, Gagner M, Urban M, Pomp A. Laparoscopic Roux-en-Y gastric bypass in patients with BMI <50: a prospective randomized trial comparing short and long limb lengths. Obes Surg. 2005 Jan;15(1):51-7. doi: 10.1381/0960892052993468. PMID 15760498
- [Background] Torres JC. Why I Prefer Gastric Bypass Distal Roux-en-Y Gastroileostomy. Obes Surg. 1991 Jun;1(2):189-194. doi: 10.1381/096089291765561268. PMID 10775917
- [Background] Fox SR, Fox KS, Oh KH. The Gastric Bypass for Failed Bariatric Surgical Procedures. Obes Surg. 1996 Apr;6(2):145-150. doi: 10.1381/096089296765557097. PMID 10729855
- [Background] Sugerman HJ, Kellum JM, DeMaria EJ. Conversion of proximal to distal gastric bypass for failed gastric bypass for superobesity. J Gastrointest Surg. 1997 Nov-Dec;1(6):517-24; discussion 524-6. doi: 10.1016/s1091-255x(97)80067-4. PMID 9834387
- [Background] Fobi MA, Lee H, Igwe D Jr, Felahy B, James E, Stanczyk M, Tambi J, Eyong P. Revision of failed gastric bypass to distal Roux-en-Y gastric bypass: a review of 65 cases. Obes Surg. 2001 Apr;11(2):190-5. doi: 10.1381/096089201321577866. PMID 11355025
- [Background] Sapala JA, Wood MH, Sapala MA, Schuhknecht MP, Flake TM Jr. The micropouch gastric bypass: technical considerations in primary and revisionary operations. Obes Surg. 2001 Feb;11(1):3-17. doi: 10.1381/096089201321454042. PMID 11361165
- [Background] Brolin RE, Cody RP. Adding malabsorption for weight loss failure after gastric bypass. Surg Endosc. 2007 Nov;21(11):1924-6. doi: 10.1007/s00464-007-9542-z. Epub 2007 Sep 3. PMID 17768659
- [Background] Pareja JC, Pilla VF, Callejas-Neto F, Coelho-Neto Jde S, Chaim EA, Magro DO. [Gastric bypass Roux-en-Y gastrojejunostomy--conversion to distal gastrojejunoileostomy for weight loss failure--experience in 41 patients]. Arq Gastroenterol. 2005 Oct-Dec;42(4):196-200. doi: 10.1590/s0004-28032005000400002. Epub 2006 Jan 19. Portuguese. PMID 16444372
- [Background] Faintuch J, Matsuda M, Cruz ME, Silva MM, Teivelis MP, Garrido AB Jr, Gama-Rodrigues JJ. Severe protein-calorie malnutrition after bariatric procedures. Obes Surg. 2004 Feb;14(2):175-81. doi: 10.1381/096089204322857528. PMID 15018745
- [Background] Spaulding L, Osler T, Patlak J. Long-term results of sclerotherapy for dilated gastrojejunostomy after gastric bypass. Surg Obes Relat Dis. 2007 Nov-Dec;3(6):623-6. doi: 10.1016/j.soard.2007.07.009. Epub 2007 Oct 23. PMID 17936088
- [Background] Mikami D, Needleman B, Narula V, Durant J, Melvin WS. Natural orifice surgery: initial US experience utilizing the StomaphyX device to reduce gastric pouches after Roux-en-Y gastric bypass. Surg Endosc. 2010 Jan;24(1):223-8. doi: 10.1007/s00464-009-0640-y. Epub 2009 Jul 25. PMID 19633885
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Deitel M, Greenstein RJ. Recommendations for reporting weight loss. Obes Surg. 2003 Apr;13(2):159-60. doi: 10.1381/096089203764467117. No abstract available. PMID 12760387
- [Background] Oria HE, Moorehead MK. Updated Bariatric Analysis and Reporting Outcome System (BAROS). Surg Obes Relat Dis. 2009 Jan-Feb;5(1):60-6. doi: 10.1016/j.soard.2008.10.004. Epub 2008 Nov 1. PMID 19161935
- [Background] Majani G, Pierobon A, Giardini A, et al. Satisfaction Profile (SAT-P) in 732 patients: focus on subjectivity in HRQoL assessment. Psychol Health 2000;15:409-22.
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery